CLINICAL TRIAL: NCT05340192
Title: Effect of Octreotide on Saliva
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00100579
Record Dates: First submitted 2022-04-15; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Healthy
MeSH Terms: interventions — Octreotide

STUDY DESIGN:
Intervention Model Description: This is a healthy volunteer pilot study. Subjects will be asked to provide a saliva sample after a 2 hour fast and 5 minutes after rinsing their mouth with tap water. The sample will be collected in an Eppendorf vial. After providing the saliva sample, each subject will be injected subcutaneously with 100 mcg (1 ml) of Octreotide by either a physician or registered nurse. A second sample of saliva will be collected using the same protocol 45-55 minutes after administering the drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Healthy Volunteer (Other): Octreotide, 100 mcg (1 ml) s.c.
  Interventions: Drug: Octreotide 1 MG/ML

INTERVENTIONS:
Drug: Octreotide 1 MG/ML — 100 mcg (1 ml) of Octreotide

SUMMARY:
The purpose of this study is to determine the effect of Octreotide on saliva enzymes. The study team hypothesizes that Octreotide will decrease the levels of certain proteins, specifically the metalloproteinase family.

DETAILED DESCRIPTION:
This is a healthy volunteer pilot study. The purpose of this study is to determine the effect of a drug, Octreotide, on saliva enzymes in order to see if this drug can help prevent pharyngo-cutaneous fistulas (an abnormal tissue connection in the pharynx) in patients undergoing laryngectomy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults between the ages of 18-40 years old
* Healthy volunteer who is willing to undergo research activities
* Healthy volunteer with no self-report of disease, oral symptoms or lesions, or cold or flu like symptoms that would affect the reflective measurements in the oral cavity
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Pregnant or nursing women
* Children under the age of 18 or adults over 40
* Complaint of oral symptoms (self-reported)
* Medical condition affecting saliva (e.g. Sjogren's)
* History of head/neck radiation
* Medication that might affect saliva (e.g. Proton Pump Inhibitors)
* Known allergy to Octreotide
* Non-English speaking
* Diabetes, gallbladder disease, heart disease, high blood pressure, a heart rhythm disorder, thyroid problems, pancreatitis, kidney disease, or liver disease (self-reported)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
To quantify the change of saliva proteomes of subjects pre-octreotide treatment | Day 1 pre-treatment
  Saliva samples analyzed using quantitative LC/MS/MS using a nanAcquity UPLC system (Waters Corp) coupled to a Thermo Orbitrap Fusion Lumos high resolution accurate mass tandem mass spectrometer (Thermo) via a nanoelectrospray ionization source
To quantify the change of saliva proteomes of subjects post-octreotide treatment | Day 1 post-treatment
  Saliva samples analyzed using quantitative LC/MS/MS using a nanAcquity UPLC system (Waters Corp) coupled to a Thermo Orbitrap Fusion Lumos high resolution accurate mass tandem mass spectrometer (Thermo) via a nanoelectrospray ionization source

CONTACTS AND LOCATIONS:
Overall Officials: Walter Lee, MD, MHS, Principal Investigator — Duke Health
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No